CLINICAL TRIAL: NCT05470257
Title: Randomized Control Trial: Elbow Extension Versus Flexion Cast in Proximal Half Both Bone Forearm Fractures
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Philip Ashley, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BBFARCT; T35HL007473 (NIH)
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Fracture of Radius and Ulna
Keywords: both bone forearm fracture; cast; pediatric
MeSH Terms: conditions — Radius Fractures | interventions — POLR1G protein, human

STUDY DESIGN:
Intervention Model Description: Two cohorts will be established. One will include patients casted in elbow extension. The other cohort will include patients casted in elbow flexion.
Masking Description: Casting is an external treatment that cannot be masked from investigators or participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elbow Flexion Cast (Experimental): This cohort will be placed in a long arm flexion cast.
  Interventions: Other: Cast
- Elbow Extension Cast (Experimental): This cohort will be placed in a long arm extension cast.
  Interventions: Other: Cast

INTERVENTIONS:
Other: Cast — Application of fiberglass long arm cast.

SUMMARY:
The purpose of this study is to compare outcomes between two immobilization methods for pediatric proximal half both bone forearm fractures.

DETAILED DESCRIPTION:
After being informed of the study including potential risks and benefits, all patients giving assent and guardian/parents consent who meet eligibility will undergo randomization of the casting technique used (elbow extension or elbow flexion casting). Randomization will occur using a random umber generator. Even numbers generated will result in an extension cast and odd numbers generated will result in a flexion cast.

The patients will be followed in clinic with an examination and x-rays at 2, 3, 5, and 8 weeks after casting to evaluate alignment of the fracture maintained by each cast. The two cohorts will be compared at the end of the study to determine which casting technique is the superior immobilization for pediatric proximal half both bone forearm fractures.

ELIGIBILITY:
Inclusion Criteria:

* Ages 3-18
* Skeletally immature
* Unilateral Radius and Ulna Fracture located within the proximal ½ of each bone
* Fracture requires reduction and casting

Exclusion Criteria:

* Ages < 3
* Distal ½ Radius and Ulna Forearm Fracture
* Isolated radius or ulna fracture
* Humerus Fracture of the Ipsilateral Arm (including floating elbow)
* Metabolic Bone Disease
* Open Fractures
* Monteggia and Galeazzi Fractures
* Deformity or abnormality not allowing for standard casting (limb deficiency, contracture)
* Parent speaks language other than english

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Alignment/Loss of Reduction | This will be accessed in clinic via x-rays until 8 weeks status post cast application.
  During clinic visits, xrays will be obtained to measure alignment of the radius and ulna fracture and asses for loss of reduction or malalignment. We will compare the number of patients with proximal both bone forearm fractures that have lost alignment after 8 weeks between the flexion elbow cast cohort compared to the extension elbow cast cohort.

SECONDARY OUTCOMES:
Cast Complications | Casting complications will be followed the full duration of the patient wearing a cast, which is expected to be around 6-8 weeks.
  We will compare the casting complications between elbow extension versus elbow flexion casting cohorts. Casting complications we will observe will be cast saw burns, cast slipping, and need for bivalve of casts.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's of Alabama, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No